CLINICAL TRIAL: NCT05747313
Title: A Prospective, Single-arm, Open-lable, Single-center Phase Ib/II Clinical Study of Chidamide in Combination With Vincristine Metronomic Chemotherapy for Advanced Triple-negative Breast Cancer
Brief Title: Chidamide in Combination With Vincristine Metronomic Chemotherapy for Advanced Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-C39
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Chemotherapy Effect
Keywords: Breast Cancer; metronomic treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Intervention Model Description: The experiment was a single-arm study design. The study is divided into two phases.
  Phase I : single-arm, open, dose-climbing Phase Ib clinical study to determine the safety and tolerability of the combination regimen and to define the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) or recommended dose for Phase II studies of this combination regimen.
  Phase II : Single-arm, open, single-center Phase II clinical study to assess the efficacy and safety of the recommended dose administered in Phase II.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Phase Ib:
  The dose of vincristine administered in this phase is 40 mg on days 1,3,5 of each cycle.
  The timepoint for chidamide dosing in this phase is twice weekly, i.e., dosing on days 1,4,8,11,15,18 of each cycle. Take 30 minutes after a meal.
  Phase II:
  This phase is based on the MTD/RP2D determined in phase I. The phase II expansion group study was conducted. Vincristine is administered at a dose of 40 mg on days 1,3,5 of each cycle. Chidamide was administered at a dose of MTD/RP2D twice a week on days 1,4,8,11,15 and 18 of each cycle. It is to be taken 30 minutes after a meal.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Phase Ib:
  The dose of vincristine administered in this phase is 40 mg on days 1,3,5 of each cycle.
  The timepoint for chidamide dosing in this phase is twice weekly, i.e., dosing on days 1,4,8,11,15,18 of each cycle. Take 30 minutes after a meal.
  Phase II:
  This phase is based on the MTD/RP2D determined in phase I. The phase II expansion group study was conducted. Vincristine is administered at a dose of 40 mg on days 1,3,5 of each cycle. Chidamide was administered at a dose of MTD/RP2D twice a week on days 1,4,8,11,15 and 18 of each cycle. It is to be taken 30 minutes after a meal.
  Other Names: Epidaza

SUMMARY:
The mechanism of action of cidabenamide and the advantages of vincristine metronomic chemotherapy make it possible to combine the two drugs. Therefore, it is necessary to conduct a prospective study to investigate the value of chidamide in combination with vincristine metronomic treatment for triple-negative breast cancer.

DETAILED DESCRIPTION:
The mechanism of action of cidabenamide and the advantages of vincristine metronomic chemotherapy make it possible to combine the two drugs. Therefore, it is necessary to conduct a prospective study to investigate the value of chidamide in combination with vincristine metronomic treatment for triple-negative breast cancer.The current study was designed to explore the efficacy of oral two-metronomic agents (chidamide in combination with vincristine) in advanced triple-negative patient in China.

ELIGIBILITY:
Inclusion Criteria:

* female;
* aged ≥ 18 years and ≤75 years;
* histologically proved metastatic triple-negative breast cancer;
* at least one measurable or evaluable lesion based on RECIST 1.1 criteria;
* estimated life expectancy ≥ 3 months; (6) normal heart, liver, and kidney function;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1; -
* informed consent signed by the participants.

Exclusion Criteria:

* received neoadjuvant or adjuvant therapy containing vinorelbine or capecitabine within one year prior to treatment initiation;
* participated in other new drug clinical trials within 4 weeks before enrollment;
* inflammatory breast cancer;
* symptomatic visceral disease;
* second primary malignancy;
* mental disorder.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | At 1 year
  1-year progression-free survival (PFS1). Evidence of local recurrence, distant metastasis, or death from any cause within 1 year counted as events in the time-to-event Kaplan-Meier analysis of progression-free survival. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions

SECONDARY OUTCOMES:
Number of Patients With Clinical Responses (Phase I) | Up to 1 year
  The number of patients with clinical responses (CR, VGPR, PR, or minimal response [MR]) will be summarized by stage.
Overall Toxicity Rate | Up to 1 year
  The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below by stage for Phase I patients.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Study Director — National Cancer Center/National Clinical Research Center for Cancer
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The individual data will not be made available in order to protect the participant's identity.